## **Borderline Personality Disorder and Emotion Regulation**

Effects of emotion-focused vs. cognitive schema therapy interventions on emotion regulation deficits in borderline personality disorder - associations between clinical efficacy, brain network function and local glutamate/GABA metabolism

Ethiks approval 04.06.2018, last time edited

## Study design



**Figure** study design: T0/T1 First therapeutic phase is divided into an active (ST-EF) and a passive (ST-AC) condition in terms of emotion-focused interventions of ST. It enables the assessment of differential effects of the experiential therapeutic techniques of ST: (i) as compared to the cognitive behavioral techniques serving as control condition (T0/T1), (ii) as compared to the influence of time (T1 vs. T2 in healthy controls), (iii) and as compared to long-term treatment effects. Marked in grey: Target group sizes as derived from the power calculation, and including possible dropouts in each group.